CLINICAL TRIAL: NCT01342666
Title: Effect of Tomato Consumption on Serum High Density Lipoprotein-cholesterol Levels. A Randomized, Open-label, Single Blind, Clinical Trial
Brief Title: Tomato Consumption and High Density Lipoprotein-cholesterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Daniel Cuevas-Ramos, MD, PhD, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REF2039
Record Dates: First submitted 2011-04-26; First posted 2011-04-27 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Hypoalphalipoproteinemia
Keywords: High density lipoprotein cholesterol; Tomato; Lycopene; Hypoalphalipoproteinemia; Dyslipidemia
MeSH Terms: conditions — Hypoalphalipoproteinemias; Dyslipidemias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tomato consumption (Experimental): Daily consumption of 300g of uncooked roma tomatoes during one month.
  Interventions: Dietary Supplement: Tomato consumption
- Cucumber consumption (Placebo Comparator): Daily consumption of 300g of cucumber.
  Interventions: Dietary Supplement: Cucumber consumption

INTERVENTIONS:
Dietary Supplement: Tomato consumption — Daily consumption of 300g of uncooked roma tomatoes during one month.
  Arms: Tomato consumption
Dietary Supplement: Cucumber consumption — Daily consumption of 300g of cucumber.
  Arms: Cucumber consumption

SUMMARY:
* This is a randomized, open-label, single blind, clinical trial
* The study evaluated the effect of tomato consumption in serum HDL-cholesterol levels.
* The hypothesis was that two daily tomatoes during one month will increase the HDL-c levels.
* Since a placebo of tomatoes cannot be done, the control group will receive same proportion of cucumber because 1) it was not possible to have a tomato placebo; 2) cucumber does not have any lycopene; 3) both can be prepared similarly; and 4) the required quantity can be measured in the same way.
* The intervention was during 1 month and was assigned by randomization.
* Personnel who did the clinical and biochemical evaluation were blinded for the intervention.
* Lipid profile was measured before and after the intervention.
* Confounding factors such as daily physical activity, diet, consumption of fish or alcoholic beverages, smoking status were considered during statistical analyses.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a main cause of death worldwide (1) and there are well recognized risk factors associated with its development. Low high density lipoprotein-cholesterol (HDL-c) rank among the most common lipid abnormalities associated with CVD (2). Low HDL-c is currently defined as an HDL-c value below 40 mg/dL for men and below 50 mg/dL for women (3). Factors related with low HDL-c are cigarette smoking (4), high triglycerides (5), sedentary lifestyle (6), and insulin resistance (7). Non-pharmacologic strategies to increase HDL-c concentration are increasing alcohol (8) and fish consumption (9), weight reduction (3), increment in physical activity (10), and smoking cessation (8). Some of these strategies are not applicable or hard to implement in individuals affected with low HDL-c. Moreover, in low-income countries, these interventions could be costly for the general population. Vegetables consumption could be a more affordable and accessible option to treat low HDL-c. Epidemiologic evidence indicates that high consumption of vegetables reduces the risk of cardiovascular disease (11) and particular attention has received tomato-based products. Growing evidence from several epidemiological studies has indicated that lycopene, the major carotenoid in tomato (12), might be more important than other carotenoids in preventing atherosclerosis and CVD (13, 14). The consumption of more than 7 servings per week of tomato-based products has been associated with a 30% reduction in the relative risk of CVD (15). Such potential benefits to vascular health from a tomato-rich diet could be related to low arterial intimal wall thickness (13, 16), reduction of LDL cholesterol levels (17), and inverse correlation with markers of inflammation and vascular endothelial dysfunction (18). However, HDL-c levels could also be positively influenced by tomato consumption. In a pilot study we found that tomato juice consumption did not increase HDL-c after one month (unpublished data), this finding also was recently reported by another group (19). In contrast, other study showed that daily consumption of 300g of uncooked tomatoes, during one month significantly increased HDL-c levels by 15.2% (20). However, this study was not controlled, not blinded, and neither randomized. Roma tomatoes consumption could be an accessible intervention to improve HDL-c levels; however, a longitudinal clinical trial is necessary to evaluate this association. Therefore, we performed a randomized, open-label, single blind, clinical trial to specifically evaluate if consumption of two uncooked tomatoes per day (14 servings/week) during one month could produce a favorable effect on HDL-c.

ELIGIBILITY:
Inclusion Criteria:

* Males with HDL-c less than 40 mg/dl
* Females with HDL-c less than 50 mg/dl
* Age between 18 to 65 years old
* Acceptance for participation with signed informed consent

Exclusion Criteria:

Previous diagnosis of:

* Diabetes,
* Hypertension,
* Kidney, liver or heart insufficiency,
* Hyperuricemia,
* Hyperandrogenic anovulation,
* Thyroid dysfunction (hypo or hyperthyroidism),
* Any difficulty to swallow appropriately, or
* Hospitalization in the previous six months.

Additionally, those subjects under current treatment with fibrates, statins, nicotinic acid, steroids, allopurinol, hormone replacement therapy (testosterone, estrogens or progesterone), metformin, other oral hypoglycemic agents, insulin, sibutramine, or orlistat treatment and those with daily consumption of any non-steroidal anti-inflammatory drug were also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Gomez-Perez, MD, FACE, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, México, Tlalpan, Mexico

REFERENCES:
- [Background] Ali MM, Agha FG. Amelioration of streptozotocin-induced diabetes mellitus, oxidative stress and dyslipidemia in rats by tomato extract lycopene. Scand J Clin Lab Invest. 2009;69(3):371-9. doi: 10.1080/00365510802658473. PMID 19148834
- [Background] Agarwal S, Rao AV. Tomato lycopene and low density lipoprotein oxidation: a human dietary intervention study. Lipids. 1998 Oct;33(10):981-4. doi: 10.1007/s11745-998-0295-6. PMID 9832077
- [Background] Arab L, Steck S. Lycopene and cardiovascular disease. Am J Clin Nutr. 2000 Jun;71(6 Suppl):1691S-5S; discussion 1696S-7S. doi: 10.1093/ajcn/71.6.1691S. PMID 10837319
- [Background] Blum A, Merei M, Karem A, Blum N, Ben-Arzi S, Wirsansky I, Khazim K. Effects of tomatoes on the lipid profile. Clin Invest Med. 2006 Oct;29(5):298-300. PMID 17144439
- [Background] Denniss SG, Haffner TD, Kroetsch JT, Davidson SR, Rush JW, Hughson RL. Effect of short-term lycopene supplementation and postprandial dyslipidemia on plasma antioxidants and biomarkers of endothelial health in young, healthy individuals. Vasc Health Risk Manag. 2008;4(1):213-22. doi: 10.2147/vhrm.2008.04.01.213. PMID 18629373
- [Background] Ashen MD, Blumenthal RS. Clinical practice. Low HDL cholesterol levels. N Engl J Med. 2005 Sep 22;353(12):1252-60. doi: 10.1056/NEJMcp044370. No abstract available. PMID 16177251
- [Background] Fuhrman B, Elis A, Aviram M. Hypocholesterolemic effect of lycopene and beta-carotene is related to suppression of cholesterol synthesis and augmentation of LDL receptor activity in macrophages. Biochem Biophys Res Commun. 1997 Apr 28;233(3):658-62. doi: 10.1006/bbrc.1997.6520. PMID 9168909
- [Background] Gianetti J, Pedrinelli R, Petrucci R, Lazzerini G, De Caterina M, Bellomo G, De Caterina R. Inverse association between carotid intima-media thickness and the antioxidant lycopene in atherosclerosis. Am Heart J. 2002 Mar;143(3):467-74. doi: 10.1067/mhj.2002.120776. PMID 11868053
- [Background] Kohlmeier L, Kark JD, Gomez-Gracia E, Martin BC, Steck SE, Kardinaal AF, Ringstad J, Thamm M, Masaev V, Riemersma R, Martin-Moreno JM, Huttunen JK, Kok FJ. Lycopene and myocardial infarction risk in the EURAMIC Study. Am J Epidemiol. 1997 Oct 15;146(8):618-26. doi: 10.1093/oxfordjournals.aje.a009327. PMID 9345115
- [Background] Re R, Mishra GD, Thane CW, Bates CJ. Tomato consumption and plasma lycopene concentration in people aged 65 y and over in a British national survey. Eur J Clin Nutr. 2003 Dec;57(12):1545-54. doi: 10.1038/sj.ejcn.1601723. PMID 14647219

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 1st of March of 2009 to 30 of April of 2011 we invited workers and patients from the INCMNSZ to participate in the study. Interested subjects were selected in a consecutive basis.
Pre-assignment Details: We performed clinical, nutritional, anthropometric, and biochemical evaluations. The protocol included a two-week run-in period with prescription of an isocaloric diet. Participants were instructed to minimize changes in diet, daily activities, specifically physical activity and smoking.
Groups:
- Tomato Consumption: Participants were randomized to receive 300 g of uncooked tomato (2 daily roma tomatoes approximately).
- Cucumber Consumption: Participants were randomized to receive 300 g of cucumber (control group).
Period: Overall Study
Arm/Group | Tomato Consumption | Cucumber Consumption
Started | 26 | 24
Completed | 26 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tomato Consumption | Cucumber Consumption | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 24 | 50
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43.4 (15.5) | 40.3 (16.0) | 41.8 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  Mexico | 26 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: High Density Lipoprotein Cholesterol (HDL-c)
Description: To evaluate the effect of two daily tomatoes consumption on HDL-c levels.
Time Frame: Baseline and after one month
Population: The sample size was calculated using the formula for means for two-tailed comparisons. According to a previous report, we expected a minimal change of 5 mg/dL in HDL-c after one month of consumption. Using a SD of 9 mg/dL with alfa of 0.05 and study power of 80%, a total of 48 subjects were calculated.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tomato Consumption | Cucumber Consumption
Number analyzed (Participants) | 26 | 24
mg/dL
  Baseline HDL-c | 36.5 (7.5) | 36.8 (7.2)
  Final HDL-c | 41.6 (6.9) | 35.8 (7.3)
Statistical Analysis 1: Comparison: Tomato Consumption vs Cucumber Consumption; We test the effect of two daily roma tomatoes during one month in HDL-c levels. We estimate the sample size to have a 80% study power; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — We did only one comparison. The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = 5.1154, 95% CI 2-sided [3.2925 to 6.9383], Standard Error of Mean 0.90570 — We compare de mean difference of the delta (final-basal levels) between groups. The values posted are the difference found in the tomato group in comparison of the control group. The mean represent the increment of HDL-c in the tomato group
Statistical Analysis 2: Comparison: Tomato Consumption vs Cucumber Consumption; Test type: Superiority or Other; p < 0.0001, Regression, Linear — A priori p value of <0.05; Adjusted for adherence, smoking, age, gender, waist to hip ratio, triglycerides, body mass index, exercise, omega 3, alcohol, fish, simple sugars; Slope = 5.656, 95% CI 2-sided [4.027 to 7.232], Standard Error of Mean 0.789 — Parameters of the model: F= 4.06; r = 0.798; r2 = 0.638; p=0.001

ADVERSE EVENTS:
Time Frame: One month, two weeks
Arm/Group | Tomato Consumption | Cucumber Consumption
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No